CLINICAL TRIAL: NCT05814575
Title: Community-based Fetal Ultrasound and Care Navigation: An Approach to Engaging Pregnant Women With Substance Use Disorder in Prenatal Care and Substance Use Treatment
Brief Title: NEXUS - Next Generation Health Through 2D & 3D Fetal UltraSound; Building Connections to Support Maternal-fetal Health
Acronym: NEXUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Principal Investigator, Amy Salisbury, Professor and Associate Dean for Research, Virginia Commonwealth University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HM20025280
Record Dates: First submitted 2023-03-03; First posted 2023-04-18 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-09

CONDITIONS: Pregnancy Related; Substance Use; Mental Health Issue
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comparator (Active Comparator): Standardized non-diagnostic fetal ultrasound protocol without interactive intervention to control for time and attention.
  Interventions: Behavioral: Standardized Non-Medical fetal ultrasound
- NEXUS Intervention (Experimental): Standardized non-diagnostic fetal ultrasound with motivational interviewing techniques, focused on maternal and fetal strengths.
  Interventions: Behavioral: NEXUS intervention; Behavioral: Standardized Non-Medical fetal ultrasound

INTERVENTIONS:
Behavioral: NEXUS intervention — During the fetal ultrasound protocol, the NEXUS intervention is added for the component of 'attachment promotion' as it is a natural extension to share with the pregnant person the behavioral and social strengths of their unborn child. As the participant observes the fetus on the monitor (a second external monitor is set up for easy viewing by the mother), she may also feel fetal movement simultaneously in the womb (after 23 weeks gestation), creating a visual and sensory link between the mother and fetus. A trained nurse or ultrasonographer shares observations of fetal behavior with the mother and others if present. The nurse is also trained in motivational interviewing techniques to use the strengths of the mother and those attributed to her fetus to explore readiness to change and other motivational factors that may be barriers to health promotion.
  Arms: NEXUS Intervention
Behavioral: Standardized Non-Medical fetal ultrasound — A standardized protocol using non-diagnostic fetal ultrasound that includes basic maternal-fetal health assessment by a trained nurse, fetal neurobehavioral assessment, measures of fetal growth, and pictures & videos given to parents.

SUMMARY:
This exploratory study brings together an interprofessional team, novel tools, and innovative, community-driven care delivery approaches to improve health equity among mother-infant dyads impacted by substance use disorder and high risk for poor health outcomes. This study will test a community-informed and community-based intervention using a fetal ultrasound protocol, motivational interviewing techniques, strength-based education, and healthcare coordination strategies to reduce health disparities faced by women and their children.

DETAILED DESCRIPTION:
Engaging women earlier in pregnancy through innovative, yet sustainable methods, will improve consistency in prenatal care and substance use treatment which will translate into substantially improved maternal and infant outcomes. The overarching premise is that successful engagement of women in accessible care during pregnancy will lead to earlier and more sustained prenatal care and treatment and lower risk for poor outcomes. This study is a multi-pronged approach to offer: (1) community-informed and community-located protocols to engage individuals into prenatal care as early as possible; (2) a novel fetal ultrasound protocol to enhance maternal-fetal connection and stimulate motivation for self-management and prenatal care; and, (3) navigation and care coordination, to connect individuals to personalized services and treatment. The NEXUS intervention is based on the idea that visualizing the fetus and seeing behavioral patterns in-utero will increase a person's sense of attachment to the fetus and in turn increase motivation for self-care and avoidance of risky behaviors. The NEXUS protocol includes a standardized fetal neurobehavioral assessment, measures of fetal growth, and, importantly, a component of 'attachment promotion' as it is a natural extension to share with the pregnant person the behavioral and social strengths of their unborn child. As the woman observes the fetus on the monitor (a second external monitor is set up for easy viewing by the mother), she may also feel fetal movement simultaneously in the womb (after 23 weeks gestation), creating a visual and sensory link between the mother and fetus. A trained nurse or ultrasonographer shares observations of fetal behavior with the mother and others if present. The family is given pictures and videos of the infant to take home with them. The NEXUS protocol will be repeated approximately 4 weeks after the first session, with educational content focused on the development of the fetus, changes in physical function, behaviors, and growth.

This is a small community-based randomized control trial in which 60 pregnant women with substance use disorder (or treatment for substance use disorder) will be offered two prenatal study visits, between the 2nd and 3rd trimesters, with two follow-up visits in the first 4 months after infant delivery. Participants will be recruited from communities with high health disparities and randomly assigned to either: (1) the Comparator Group which receives a standard non-diagnostic ultrasound with minimal interaction and no accompanying education or, (2) NEXUS Intervention Group which receives the NEXUS fetal ultrasound protocol that includes motivational interviewing and content specific to emotional and cognitive connection with the fetus. The prenatal ultrasound visits and the follow-up visits will be offered within the community in which the participant lives. All participants will receive standardized education, care coordination, and weekly contact with care navigators.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant persons, Aged 18 through 45, between 22-32 weeks gestation at study entry
* Provision of signed and dated informed consent form
* Not incarcerated
* Able to read and understand English
* For infants after delivery, parental informed consent to participate in the study
* Stated willingness to comply with all study procedures
* Meets Diagnostic and Statistical Manual 5 criteria for Substance Abuse or substance use disorder in the last 12 months or is in active treatment for substance use disorder (including Nicotine/Tobacco, alcohol, marijuana, illicit and licit substances, and opioids) or actively using substances during pregnancy.
* Willingness to participate in the NEXUS regimen

Exclusion Criteria:

* Presenting with cognitive impairment
* psychiatric instability (active psychosis or acute mania)
* language or legal barriers that would limit the patient's ability to provide informed consent and complete research assessments.
* Known fetal anomalies
* Medical conditions requiring frequent ultrasound monitoring outside the study (e.g.

Gestational Diabetes)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 103 (Actual)
Dates: Start 2023-06-08 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Study Retention | 10-26 weeks
  Percentage of each group returning for a second study visit
Parent Subjective Connection to Fetus/Infant | Baseline through 12 Weeks post-delivery
  Participants reported scores of maternal-fetal attachment at the Baseline visit and at last postpartum session; Maternal-fetal attachment scale; Parent-Infant Attachment Questionnaire at 12 weeks post-delivery; (0-5 score, higher is better)
Prenatal care utilization | Immediately following infant birth
  The number of prenatal care visits per week of gestation at delivery.
Substance use treatment utilization | Immediately following infant birth
  The number of substance use and mental health treatment visits per week of gestation at delivery.

SECONDARY OUTCOMES:
Access to Care | 26 weeks
  PRAMS access to care survey
Perceived Stress | 26 weeks
  Perceived Stress Scale
Substance use in pregnancy | Immediately following infant birth
  Participants' reported substance use at weekly check-ins during and after pregnancy: total number of days using substances in pregnancy (tobacco, alcohol, illicit drugs, marijuana).
Obstetric complications | 12 weeks postpartum
  The total number of Obstetrics Complications identified by participant reports and medical record occurring from pregnancy through 12 weeks postpartum.

CONTACTS AND LOCATIONS:
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized participant data will be shared in a standard data repository.
Supporting Information: Study Protocol, SAP
Time Frame: To be determined
Access Criteria: To be determined

DOCUMENTS (1):
  • Informed Consent Form (2024-04-25): https://cdn.clinicaltrials.gov/large-docs/75/NCT05814575/ICF_000.pdf